CLINICAL TRIAL: NCT06136065
Title: 68Ga-FAPI-46 Positron Emission Tomography - Computerized Tomography for Molecular Assessment of Fibroblast Activation
Brief Title: 68 Gallium-Fibroblast Activating Protein Inhibitors-46 Positron Emission Tomography - Computerized Tomography for Molecular Assessment of Fibroblast Activation and Risk Assessment in Solid Tumors
Acronym: FAPI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRST 100.59; 2022-003786-38 (EudraCT Number); 2024-511659-17-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-13; First posted 2023-11-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor, Unspecified, Adult
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: A total of 100 patients will be enrolled. The proportion of 68-Gallium-Fibroblast Activating Protein Inhibitor-46 Positron Emission Tomography /Computerized Tomography positive patients or lesions will be calculated as well as 95% confidence intervals (CI). Median and ranges or mean and standard deviation, as appropriate, will be used to describe 68-Gallium-Fibroblast Activating Protein Inhibitor-46 (68Ga-FAPI-46) uptake. The number and percentage of treated patients undergoing grade 1 to 4 adverse events will be tabulated according to CTCAE version 5.0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): 100 patients with solid tumor and 18-Fluorine-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose Positron emission tomography / Computerized tomography scan dubious
  Interventions: Diagnostic Test: 68 Gallium -Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography

INTERVENTIONS:
Diagnostic Test: 68 Gallium -Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography — 68 Gallium -Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography scan

SUMMARY:
Phase II, open label, single arm, single center, prospective diagnostic trial to evaluate the Fibroblast Activating Protein (FAP) positivity in patients with solid tumors

DETAILED DESCRIPTION:
The growth and spread of the tumor is determined not only by the tumor cells but also by the non-malignant constituents of the malignant lesion, which contributes to what is commonly referred to as the "tumor microenvironment". In particular, a subpopulation of fibroblasts called cancer-associated fibroblasts are involved in tumor growth, migration and progression. Therefore, these cells represent an attractive target for both diagnosis and anticancer therapy.

A distinctive feature of cancer-associated fibroblasts is the expression of the fibroblast activating protein, a type II membrane-bound glycoprotein. Fibroblast Activating Protein plays a role in normal developmental processes during embryogenesis and in tissues modeling.

The presence of Fibroblast Activating Protein in cancer-associated fibroblasts in many solid tumors and the fact that overexpression is associated with a worse prognosis in cancer patients has led to the hypothesis that Fibroblast Activating Protein plays a fundamental role in the development of cancer, in the migration of cancer cells, and in the spread of cancer. Therefore, the targeting of this enzyme for imaging and endo-radiotherapy can be seen as a promising strategy for detecting and treating malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically solid tumors at any stage, if biopsy is no feasible for technical reason or risk benefit balance, patients may be enrolled if CT or MRI strongly suggest oncological lesion;
2. 18-Fluorine-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose Positron emission tomography / Computerized tomography or other clinical practice morpho-functional imaging scan dubious or inconclusive;
3. Male or Female, aged>18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status <2 (see Appendix A)
5. A female participant is eligible to participate if she is not pregnant and not breastfeeding. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (See Appendix D) are mandatory. Highly effective birth control methods are required beginning at the screening visit and continuing at least 6 months following last treatment with study drug. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required ( established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg., bilateral orchiectomy), for more than 6 months.
6. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Participation in another clinical trial with any investigational agents within 30 days prior to study entry or 5 half lives of the study drug.
2. Medical or psychological conditions that would not allow the participant to understand, or sign the informed consent
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Fibroblast Activating Protein Inhibitor or other agents used in the study.
4. Inability to remain still for the entire duration of the exam
5. Life expectancy < 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance status > 2
7. Patient with compromised renal function (Creatinine> 2 mg/ml)
8. Patient with altered hepatic function (AST and Alanine Aminotransferase > 2.5 respect to upper normal limits)
9. Pregnancy and lactation
10. Subject deprived of its freedom by administrative or legal decision or who is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68-Gallium -Fibroblast Activating Protein Inhibitor - 46 Positron emission tomography / Computerized tomography | 30 months
  ratio between the number of 68 Gallium - Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography positive patients and the number of patients with solid tumors presenting with Fluorodeoxyglucose Positron Emission Tomography/Computerized Tomography scan or other clinical practice morpho-functional imaging dubious or inconclusive.

SECONDARY OUTCOMES:
Detection rate of lesions, stratified by tumor histology | 30 months
  Proportion of positive patients on total number who underwent 68 Gallium -Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography stratified for tumor histotypes
Detection rate of stratified lesions for different lesion sites | 30 months
  Proportion of positive patients on total number who underwent 68 Gallium -Fibroblast Activating Protein Inhibitor -46 Positron emission tomography / Computerized tomography stratified for different lesion sites
Uptake of 68 Gallium -Fibroblast Activating Protein Inhibitor -46 | 30 months
  Uptake of 68 Gallium - Fibroblast Activating Protein Inhibitor - 46 in terms of SUV
Safety (percentage of patients) | 30 months
  safety is defined as the percentage of treated patients undergoing grade 1 to 4 adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Istituto ROmagnolo per lo Studio dei Tumori "Dino Amadori"-IRST S.r.l., Meldola, Forlì Cesena
  - Azienda USL Toscana Centro - SOC Medicina Nucleare - Nuovo Ospedale "Santo Stefano", Prato

IPD SHARING:
Plan to Share IPD: No